CLINICAL TRIAL: NCT07363057
Title: Phase 2a, Proof-Of-Concept, Multi-National, 8-Week, Randomized, Single-Blinded, Placebo-Controlled Trial of GI-102 in Combination With GIB-7 to Evaluate Its Effects on Biomarkers of Aging in Healthy Adults and Cancer Survivors
Brief Title: A Study to Evaluate the Effects of the Combination of GI-102 With GIB-7 on Biomarkers of Aging in Healthy Adults and Cancer Survivors
Acronym: GIANTS-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GI Innovation, Inc. (Industry)
Collaborators: GILongevity (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GIANTS-1
Record Dates: First submitted 2025-12-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer Survivors; Healthy Participant; Elderly
Keywords: GI-102; GIB-7; aging; immunosenescence; gut-brain-muscle axis dysregulation; metabolic dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Active Comparator): GI-102 in combination with GIB-7
  Interventions: Combination Product: GI-102 in combination with GIB-7
- Part B Arm 1 (Active Comparator): GI-102 in combination with GIB-7
  Interventions: Combination Product: GI-102 in combination with GIB-7
- Part B Arm 2 (Placebo Comparator): Placebo for GI-102 in combination with GIB-7
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: GI-102 in combination with GIB-7 — GI-102: recombinant protein drug, intravenous (IV) infusion, once every 4 weeks (Q4W); GIB-7: synbiotic formula, oral administration, once daily (QD)
  Other Names: efzilonkofusp alfa in combination with GIB-7
  Arms: Part A; Part B Arm 1
Combination Product: Placebo — Placebo for GI-102 in combination with GIB-7
  Arms: Part B Arm 2

SUMMARY:
This Phase 2a clinical study (GIANTS-1) aims to evaluate a novel dual-combination strategy using GI-102 and GIB-7 to address key pathological features of aging, including immunosenescence (the aging of the immune system), metabolic dysfunction, and gut-brain-muscle axis dysregulation.

DETAILED DESCRIPTION:
GI-102 targets immunosenescence and inflammation: GI-102 is a bispecific immunocytokine composed of CD80 fused with a mutated interleukin (IL)-2. It is currently being evaluated in an ongoing Phase 2 oncology study, in which its safety and tolerability has been evaluated. Clinically meaningful biological activity-such as increased peripheral lymphocyte counts (including CD8+ T cells and natural killer [NK] cells)-has been observed, supporting its potential role in immune reactivation and inflammation modulation in the aging population.

GIB-7 restores gut-brain-muscle axis and circadian rhythm: GIB-7 is a proprietary synbiotic formulation that contains four probiotic strains- Limosilactobacillus fermentum, Lactiplantibacillus plantarum, which are gram-positive lactic acid bacteria. Additionally, it contains the strains Lactobacillus acidophilus, and Bifidobacterium animalis subsp. lactis. These components collectively support gut microbial stability and systemic physiological balance. In a clinical study conducted in healthy older adults (NCT05735418), GIB-7 demonstrated significant improvements in grip strength and reductions in inflammatory markers, with no investigational product (IP)-related adverse events (AEs), confirming its excellent safety profile. Additionally, GIB-7 has been shown to support circadian rhythm regulation, a key aspect of homeostatic aging that is often disrupted in older adults.

The rationale for combining these two agents is their complementary mechanisms:

* GI-102 aims to remove senescent cells and thereby reduce inflammaging (a form of low-grade inflammation associated with ageing) via immune reactivation.
* GIB-7 aims to enhance gut stability and support the gut-brain-muscle axis and circadian alignment, thereby improving physical and cognitive resilience.

This dual-combination strategy addresses complementary hallmarks of aging, offering a mechanistically integrated approach to extending healthspan (the period during which individuals remain functional and free of chronic diseases) in healthy adults and cancer survivors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must be aged between ≥18 and ≤80 years old at the time of informed consent.
2. At the discretion of the Investigator, must be in a state of general health that is not severely compromised (ie, no life-threatening illness or disability).
3. Participants with a history of cancer may be included only if they meet one of the following:

   1. Participants have been disease-free for ≥2 years; OR
   2. For those diagnosed within 2 years:

      * The cancer was treated with curative intent (eg, surgery, anti-cancer agents including chemotherapy)
      * Participants have been in remission for ≥12 months
      * Participants are not on any active cancer treatment except maintenance therapies (eg, endocrine therapy or bisphosphonates)
      * Participants must have received systemic anti-cancer therapies without immunotherapy for their cancers
4. Women of childbearing potential (WOCBP; see definition in Section 5.3) must agree to use a highly effective method of contraception from 14 days prior to Visit 2 until 180 days after the last dose of study medication (GI-102 or GIB-7). Fertile men must agree to use an acceptable method of contraception from 14 days prior to Visit 2 until 90 days after the last dose of study medication (GI-102 or GIB-7).

Key Exclusion Criteria:

1. Severe and poorly managed chronic diseases, such as advanced cardiovascular disease, kidney failure requiring transplant or dialysis, uncontrolled diabetes, detectable malignancy (≤ 2 years), severe chronic obstructive pulmonary disease (COPD), or untreatable, terminal cancer as judged by the Investigator or history of life threatening infection (eg, meningitis).
2. Dependent on walkers or wheelchairs; severe difficulty or inability to perform activities of daily living independently or inability to perform study measures required to test muscle function (an amputee is eligible if participants can walk without walkers or wheelchair) as judged by the Investigator.
3. Major surgery within the past 6 months or scheduled during the study period, including severe orthopedic diseases requiring joint replacement surgery.
4. History of substance abuse or dependency or history of recreational IV drug use over the last 5 years (by self-declaration).
5. Female participants who are pregnant, planning to become pregnant, or breastfeeding during the study period. Participants undergoing perimenopause or the menopause transition are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline values in immune response (NK cells) before and after GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Maximum change from Baseline values in immune function, primarily in natural killer (NK) cells assessed by flow cytometry in blood samples.
Change in Baseline values in immune response (CD8+ T cells) before and after GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Maximum change from Baseline values in immune function, primarily in CD8⁺ T cells assessed by flow cytometry in blood samples.
Frequency of Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) of the combination of GI-102 and GIB-7 by severity | From Day 1 until Week 10 visit
  Frequency of Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) by severity.
Number of participants with various adverse events and abnormal lab data | From Day 1 until Week 10 visit
  Number of participants with Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), abnormal Vital signs, abnormal Electrocardiograms (ECGs), abnormal Physical examination findings, abnormal Chest X-ray, or abnormal Laboratory tests results

SECONDARY OUTCOMES:
Change in Baseline values in sleep quality before and after GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Change from Baseline values in sleep quality using ISI (Insomnia Severity Index) at Week 8 and Week 10
Change in Baseline values in quality of life before and after GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Change from Baseline values in quality of life using EQ-5D (EuroQol 5 Dimension) at Week 8 and Week 10
Change in Baseline values in muscle function (hand grip strength) before and after GI-102 and GIB-7 combination treatment | From enrollment to the end of study
  Change from Baseline values in muscle function using hand grip strength test at Week 8 and Week 10
Change in Baseline values in muscle function (6 minute walk test) before and after GI-102 and GIB-7 combination treatment | From enrollment to the end of study
  Change from Baseline values in muscle function using 6 minute walk test at Week 8 and Week 10

OTHER OUTCOMES:
Change in Baseline values in the hospital visits by GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Number of hospital visits compared to placebo at Week 8 and Week 10 (falls, fractures, pneumonia or severe respiratory illness, and other major health events may also be collected) to be conducted in a subgroup analysis (≥ 50 years)
Change in Baseline values in gut microbiome by GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Change from Baseline values in gut microbiome at Week 8 and Week 10 as indicated by fecal microbiota changes using alpha-diversity values and taxonomic relative abundances.
Change in Baseline values in cognitive function by GI-102 and GIB-7 combination treatment | From Day 1 until Week 10 visit
  Change from Baseline values in cognitive function at Week 8 and Week 10 as assessed by MoCA (Montreal Cognitive Assessment)
Survival (cancer survivors only) | From Day 1 until Week 10 visit
  In this study investigators will monitor overall survival defined as time from the inclusion to death or end of follow up at Week 10 (whichever comes first).
Recurrence (cancer survivors only) | From Day 1 until Week 10 visit
  In this study investigators will monitor cancer recurrence defined as time from the inclusion to the first recurrence or end of follow up at Week 10 (whichever comes first).

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Novatrials, Charlestown, New South Wales
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Yes
Data and biospecimens collected in this study may be accessed by the XPRIZE Foundation and its designated Judging Panel solely for the purpose of verifying study results and evaluating eligibility for the XPRIZE Healthspan Competition.
  No identifiable personal information will be shared, and all data provided will remain confidential and used only for competition judging and audit purposes.